CLINICAL TRIAL: NCT07259642
Title: Clinical Comparison of Different Debonding Techniques of Clear Aligner Attachments: A Single-center, Split-Mouth Randomized Clinical Trial
Brief Title: Comparison of Different Debonding Techniques of Clear Aligner Attachments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ezgi Atik, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-22-03
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Orthodontic Pain (D013850); Orthodontic Patient Experience; Orthodontic Aligners; Orthodontic
Keywords: Debonding, clear aligner attachment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plier group (Experimental): In this group, clear aligner attachments are removed using adhesive removal pliers , followed by cleaning of residual adhesive with a 24-blade tungsten carbide finishing bur operated at low speed (20,000 rpm) without water cooling.
  Interventions: Procedure: Adhesive removal plier followed by tungsten carbide bur
- Bur Group (Active Comparator): In this group, clear aligner attachments are completely removed using a 24-blade tungsten carbide bur operated at low speed (20,000 rpm) without water cooling.
  Interventions: Procedure: Tungsten carbide bur

INTERVENTIONS:
Procedure: Adhesive removal plier followed by tungsten carbide bur — In this intervention, clear aligner attachments are removed using an adhesive removal plier with a controlled torquing motion. After mechanical detachment of the attachments, any remaining adhesive resin is removed using a 24-blade tungsten carbide finishing bur operated at low speed (20,000 rpm) without water cooling. This combined approach aims to minimize discomfort by reducing contact time with rotary instruments while ensuring complete adhesive removal. Pain levels are evaluated immediately after debonding each segment using an 11-point Numeric Rating Scale (NRS). Adhesive remnants are scored using a modified Adhesive Remnant Index (ARI) before bur refinement.
  Arms: Plier group
Procedure: Tungsten carbide bur — In this intervention, clear aligner attachments are completely removed using a 24-blade tungsten carbide bur operated at low speed (20,000 rpm) without water cooling. No plier is used in this method. Pain levels are evaluated immediately after debonding each segment using an 11-point Numeric Rating Scale (NRS). This continuous rotary technique represents a conventional clinical approach for attachment removal.
  Arms: Bur Group

SUMMARY:
The goal of this clinical trial is to compare two different methods for removing clear aligner attachments from tooth surfaces and to evaluate the pain levels and removal times associated with each method. The main questions this study aims to answer are:

* Does the use of an adhesive removal plier result in less pain compared to using a tungsten carbide bur?
* Is there a difference in the time required to remove attachments between the two methods?

In this split-mouth, randomized clinical trial, participants who have completed clear aligner treatment will undergo two different attachment removal techniques:

* Plier method: Attachments will be removed using adhesive removal pliers, followed by finishing with a tungsten carbide bur.
* Bur method: Attachments will be removed entirely using a tungsten carbide bur. Pain levels will be assessed using an 11-point Numeric Rating Scale (NRS) after each segment is treated, and the time required for each removal will be recorded. The amount of adhesive remaining on the enamel surface will also be evaluated.

This study aims to determine which debonding technique provides a faster and more comfortable experience for patients at the end of aligner treatment.

DETAILED DESCRIPTION:
This study was conducted to compare two different debonding techniques used for removing clear aligner attachments and to evaluate their effects on pain perception, removal time, and adhesive remnants on the enamel surface. Clear aligner attachments are routinely used to enhance tooth movement, and their removal at the end of treatment should be efficient, safe, and comfortable for patients. However, there is limited clinical evidence evaluating patient-centered outcomes.

This single-center, split-mouth, randomized clinical trial included participants who had completed clear aligner treatment or the first set of clear aligners and required removal of composite attachments. Each participant received both debonding techniques in diagonally opposite quadrants to allow direct comparison within the same individual. In the plier technique, attachments were mechanically disengaged using adhesive removal pliers, followed by refinement of the enamel surface with a 24-blade tungsten carbide finishing bur. In the bur technique, attachments were completely removed using a 24-blade tungsten carbide bur without prior mechanical detachment. All procedures were performed at low speed and without water cooling.

Pain intensity was assessed immediately after debonding each segment using the Numeric Rating Scale (NRS), an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable), where higher scores indicate worse pain. Removal time for each attachment was recorded using a digital timer. Adhesive remnants were evaluated using a modified Adhesive Remnant Index (ARI) scored from 0 to 2. Additional analyses examined whether pain scores differed by age, gender, and attachment type (optimized vs. conventional).

The overall aim of this study was to provide clinically relevant evidence to guide orthodontists in selecting an attachment removal technique that maximizes patient comfort, improves clinical efficiency, and minimizes adhesive remaining on the enamel surface at the end of clear aligner therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 44 years with permanent dentition
* No history of taking medication in the last 24 hours (e.g., painkillers, corticosteroids, and antiflu drugs)
* Patients with no missing teeth except for third molars
* Patients who underwent clear aligner treatment (Invisalign®) without an extraction protocol by one of the co-authors of the present study
* Patients who completed aligner treatment and reached the attachment removal stage
* Patients with at least 4 attachments in each quadrant of the mouth and a total of at least 16 attachments
* Patients in good general and oral health with no periodontal disease

Exclusion Criteria:

* Patients with endodontic treatment, large restorations, and buccal restorations
* Patients with a history of previous orthodontic treatment
* The presence of systemic diseases that may cause dentin and enamel hypersensitivity
* Patients who underwent surgical treatment and displayed signs of gingival recession
* Patients who received teeth whitening in the last 8 weeks.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain level during attachment removal | Immediately after debonding each segment
  Pain intensity will be measured immediately after debonding each segment (anterior and posterior) using an 11-point Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores indicate worse pain. In group pliers, pain levels were recorded separately after both plier and bur applications for each segment, and the average was calculated to provide a single pain value. In bur group, pain scores were recorded after each segment attachments were completely removed.

SECONDARY OUTCOMES:
Attachment removal time per tooth | Immediately after debonding each segment
  The removal time per quadrant was calculated in seconds by a digital timer. The average removal time required per attachment was calculated by dividing the total attachment removal time in each quadrant by the number of attachments present in that quadrant.
Adhesive remnants on enamel surface | Immediately after attachment removal with pliers
  In the Plier group, after debonding attachments with a plier and before removing the residual adhesive with a bur, a modified adhesive remnant index (ARI) was used to evaluate the remaining adhesives using a magnifying dental loupe at 2.5X magnification by two examiners. "0" indicated no adhesive remaining on the tooth, "1" indicated less than half of the adhesive remaining, and "2" indicated more than half remaining. Higher scores indicate more adhesive remaining. If there were discrepancies, a third examiner was asked to make the final determination of the score.
Comparison of pain levels between genders | Immediately after debonding each segment
  NRS pain scores obtained during debonding will be compared between male and female participants to evaluate potential gender-related differences in pain perception.
Correlation between age and pain perception | Immediately after debonding each segment
  The relationship between participants' age and reported NRS pain scores will be analyzed to determine whether pain perception varies by age.
Comparison of adhesive remnant index (ARI) according to attachment type (optimized vs. conventional) | Immediately after debonding using the plier technique
  After attachment removal using the plier technique, the distribution of ARI scores will be compared between optimized and conventional attachment types to determine whether attachment design influences the amount of adhesive remaining on enamel surfaces.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Atik, Dr., Principal Investigator — Hacettepe University Faculty of Dentistry Department of Orthodontics
Locations (1):
- Hacettepe University Faculty of Dentistry Department of Orthodontics, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared in order to protect participants' privacy and ensure compliance with institutional and ethical data protection regulations. All collected data contain potentially identifiable information, and therefore will remain confidential and stored securely within the study institution.